CLINICAL TRIAL: NCT05558449
Title: Impact of Virtual Reality Hypno-sedation on Functional Recovery and Anxiety in Foot Surgery With Regional Anesthesia: a Randomized Clinical Trial.
Brief Title: Impact of Virtual Reality Hypno-sedation on Functional Recovery and Anxiety in Foot Surgery With Regional Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Michele Carella, Head of Clinic, Anesthesiology and Intensive Care Department, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VRH.foot
Record Dates: First submitted 2022-09-22; First posted 2022-09-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Foot Deformities; Regional Anesthesia Morbidity; Valgus; Hallux; Analgesia
MeSH Terms: conditions — Foot Deformities; Hallux Valgus; Agnosia | interventions — Hypnosis, Anesthetic; Midazolam

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Clinical Trial
Masking Description: Open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR (Active Comparator): Patients in the VR group (19 patients) will receive VR alone without hypnosedation. The VR headset will be used on these patients without an external voice or device allowing hypnosis. The VR module used will be "Silva", i.e. a scenario of a walk in the forest through the 4 seasons.
  Interventions: Device: Virtual reality
- VRH (Experimental): The patients in the VRH group (19 patients) will benefit from a hypnosedation session with a VRH headset during the local anesthesia technique and during the surgery (approximately 60 minutes). The VRH module used will be "Silva", i.e. the same scenario of a walk in the forest through the 4 seasons with a voice accompanying the hypnosis session.
  Interventions: Device: Hypnosedation
- C (Active Comparator): Patients in group C (control group, 19 patients) will receive only midazolam-based pharmacological sedation. This will be administered with intermittent boluses of 1 mg until patient comfort and sedation on the Richmond analgo-sedation scale (RASS) of -3 (response to verbal stimulus) is achieved.
  Interventions: Drug: Midazolam injection

INTERVENTIONS:
Device: Hypnosedation — Hypnosedation session with a virtual reality headset during the regional anesthesia technique and during the surgery (approximately 60 minutes). The VRH module used will be "Silva", i.e. the same scenario of a walk in the forest through the 4 seasons with a voice accompanying the hypnosis session.
  Arms: VRH
Drug: Midazolam injection — Midazolam intravenous injection 1 mg until RASS -3
  Arms: C
Device: Virtual reality — Only virtual reality without a hypnosedation session. The virtual reality headset will be used on these patients without external voice or hypnosis device. The virtual reality module used will be "Silva", i.e. a scenario of a walk in the forest through the 4 seasons.
  Arms: VR

SUMMARY:
This prospective study aims to evaluate whether the implementation of a virtual reality hypnosedation (VRH)protocol reduces preoperative anxiety and increases patient comfort before, during, and after outpatient foot surgery.

DETAILED DESCRIPTION:
This prospective study aims to evaluate whether the implementation of a virtual reality hypnosedation (VRH) protocol reduces preoperative anxiety and increases patient comfort before, during, and after outpatient foot surgery. The investigators hope to demonstrate a reduction in anxiety, improved postoperative experience and functional recovery according to currently validated scores measuring preoperative and postoperative recovery, anxiety and stress, and experience during a regional anesthesia technique.

The investigators expect that VRH will be more effective than VR alone and conventional pharmacological sedation in reducing preoperative anxiety and in improving experience and functional recovery. If the hypothesis is correct, the investigators could propose to integrate this protocol as a first line in the ambulatory management of elective foot surgery.

ELIGIBILITY:
Inclusion Criteria:

* Major patients, classified as ASA 1-2-3, admitted for foot surgery (metatarsophalangeal arthrodesis or hallux valgus cure), under peripheral locoregional anesthesia (sciatic nerve block at popliteal level).

Exclusion Criteria:

* pregnant women
* patients with peripheral neuropathy or other severe neurological pathology
* allergy or contraindication to local anesthetics or benzodiazepines
* chronic renal failure or severe hepatic failure
* major hemostasis disorders
* severe vision or hearing problems that would render the VR and VRH device useless or unusable, and patient contraindication or refusal to use the VRH headset, such as claustrophobia or kinesiophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
(Evaluation du Vecu de l'Anesthesie LocoRegionale) EVAN-LR | 4 hours after surgery
  The primary endpoint will be the EVAN-LR score as a measure of intraoperative experience. EVAN-LR: a 0-100 scale, with 100 indicating the best possible level of satisfaction and 0 the worst.

SECONDARY OUTCOMES:
Anxiety | 5 minutes after the end of the surgery
  Numeric rating scale (NRS) (0 to 10) for pre- and postoperative anxiety
Quality of Recovery- 15 items (QoR-15) | 1 day before, 1 and 3 day after surgery
  Assessment of the QoR-15 score on postoperative functional recovery and the variation in time between the day before surgery, the day after and 3 days after surgery
Length of surgery | 5 minutes after the end of the surgery
  Length of surgery procedure in minutes
Complications | 6 hours after surgery
  The occurrence of complications related to the techniques used
VRH complications | 6 hours after surgery
  The occurrence of side effects related to virtual reality (nausea, paradoxical anxiety, dizziness, etc.)
Time perception | 5 minutes after the end of the surgery
  Perception of the duration of the surgery during the VRH.
Surgeon satisfaction | 5 minutes after the end of the surgery
  Surgeon satisfaction on a numeric rating scale from 0 to 10
Dissociation | 5 minutes after the end of the surgery
  The Numeric rating scale (NRS) (0-10) dissociation for the assessment of dissociation during the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carella M, Bicego A, Beck F, Malta C, Ardizzone L, Bonhomme VL, Vanhaudenhuyse A. Influence of virtual reality with or without hypnosis on patient-related experience and functional recovery in outpatient foot surgery with regional anesthesia: a randomized controlled trial. Reg Anesth Pain Med. 2025 Jun 22:rapm-2025-106678. doi: 10.1136/rapm-2025-106678. Online ahead of print. PMID 40545295